CLINICAL TRIAL: NCT04637295
Title: Perceptions, Experiences, and Activity in CancEr Survivors During COVID-19
Acronym: PEACE
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0768-20-EX
Record Dates: First submitted 2020-11-17; First posted 2020-11-19 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Neoplasms Malignant
Keywords: Physical Activity; COVID; Cancer
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To examine perceptions and determinants of physical activity during the COVID-19 pandemic among cancer survivors.

DETAILED DESCRIPTION:
This purpose of this study is to examine perceptions and determinants of physical activity during the COVID-19 pandemic in cancer survivors. To test our aim, we will recruit up to 1000 adults diagnosed with cancer within the last five years and ask them to complete an online questionnaire battery assessing their self-reported physical activity habits, psychosocial outcomes (e.g., depression, anxiety, self-efficacy, social support), and perceptions of physical activity engagement during the pandemic. A subsample of participants (n=50) will also be invited to participate in an interview to gain further insights into cancer survivors' physical activity experiences during COVID-19. Analysis of covariance (ANCOVA) will be used to analyze the quantitative survey data, and thematic analysis will be used to analyze the qualitative interview data.

ELIGIBILITY:
Inclusion Criteria:

* Adult with a history of cancer (except non-invasive skin cancer)
* Diagnosed at age 19 or older
* Diagnosed within 5 years of study enrollment
* Access to a computer, tablet, or smartphone with the Internet
* English reading

Exclusion Criteria:

* Unable to read in English

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruiting cancer survivors who have been diagnosed within the last 5 years. Survivors can be at any stage of their cancer diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2021-06-17 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 14 days
  Godin Leisure-Time Exercise Questionnaire
Psychosocial Function during COVID-19 | 14 days
  COVID-19 Pandemic Psychosocial Functioning Measure

SECONDARY OUTCOMES:
Self-Efficacy | 14 days
  The Exercise Self-efficacy Scale will be used to measure confidence in ability to exercise. A higher score indicated a higher confidence.
Sleep Quality | 14 days
  The Pittsburgh Sleep Quality Index will be used to measure sleep quality and disturbances. A higher score indicates a higher sleep disturbance.
Fatigue | 14 days
  The Functional Assessment in Chronic Illness Therapy - Fatigue (FACIT-F) will be used to measure fatigue as well. Higher scores indicate less fatigue.
Anxiety | 14 days
  The Hospital Anxiety and Depression Scale (HADS) will be used to produce an anxiety score. Higher scores indicate higher symptoms of anxiety.
Depression | 14 days
  The Hospital Anxiety and Depression Scale (HADS) will be used to produce an anxiety score. Higher scores indicate higher symptoms of depression.
Loneliness | 14 days
  The UCLA Loneliness Scale will be used to measure feelings of loneliness and isolation. Higher scores indicate higher degrees of loneliness.
Global Self-Esteem | 14 days
  The Rosenberg Self-Esteem Scale (RSE) will be used to measure global self-esteem. Items are used to calculate an esteem score, higher scores are indicative of higher esteem.
Subjective Cognitive Impairment | 14 days
  The Functional Assessment in Cancer Therapy- Cognition (FACT-Cog) measures levels of cognitive impairment, quality of life and perceived cognitive ability. Items are summed up to calculate scores from each subsection.
Social Support | 14 days
  The Social Support of Exercise scale is aimed to assess the degree in which family and friends demonstrate support for exercise behavior. Higher scores indicate a higher level of support.
Satisfaction of Life | 14 days
  The Satisfaction of Life Scale (SWLS) is developed to assess global satisfaction is various age groups.
Stress | 14 days
  The Perceived Stress Scale is a 10-item scale developed to measure the perceptions of a person's stress.
Perceptions of Exercise | up to one month after enrollment
  A qualitative interview will be performed to measure the perceptions and barriers of exercise during the COVID-19 pandemic. This interview is comprised of items designed by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Diane K Ehlers, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
Select data may be shared upon request of the primary investigator.

REFERENCES:
- [Background] Godin G, Shephard RJ. A simple method to assess exercise behavior in the community. Can J Appl Sport Sci. 1985 Sep;10(3):141-6. PMID 4053261
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Hoch CC, Yeager AL, Kupfer DJ. Quantification of subjective sleep quality in healthy elderly men and women using the Pittsburgh Sleep Quality Index (PSQI). Sleep. 1991 Aug;14(4):331-8. PMID 1947597
- [Background] Basen-Engquist K, Bodurka-Bevers D, Fitzgerald MA, Webster K, Cella D, Hu S, Gershenson DM. Reliability and validity of the functional assessment of cancer therapy-ovarian. J Clin Oncol. 2001 Mar 15;19(6):1809-17. doi: 10.1200/JCO.2001.19.6.1809. PMID 11251013
- [Background] Yellen SB, Cella DF, Webster K, Blendowski C, Kaplan E. Measuring fatigue and other anemia-related symptoms with the Functional Assessment of Cancer Therapy (FACT) measurement system. J Pain Symptom Manage. 1997 Feb;13(2):63-74. doi: 10.1016/s0885-3924(96)00274-6. PMID 9095563
- [Background] Snaith RP. The Hospital Anxiety And Depression Scale. Health Qual Life Outcomes. 2003 Aug 1;1:29. doi: 10.1186/1477-7525-1-29. PMID 12914662
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Robins, R. W., Hendin, H. M. & Trzesniewski, K. H. Measuring global self-esteem: Construct validation of a single-item measure and the Rosenberg Self-Esteem Scale. Personal. Soc. Psychol. Bull. 27, 151-161 (2001).
- [Background] Wagner, L. I., Sweet, J., Butt, Z., Lai, J. & Cella, D. Measuring patient self-report cognitive function: Development of the functional assessment of cancer therapy-cognitive function instrument. J. Support. Oncol. 7, W32-W39 (2009).
- [Background] Resnick B, Orwig D, Magaziner J, Wynne C. The effect of social support on exercise behavior in older adults. Clin Nurs Res. 2002 Feb;11(1):52-70. doi: 10.1177/105477380201100105. PMID 11845515
- [Background] Pavot W, Diener E, Colvin CR, Sandvik E. Further validation of the Satisfaction with Life Scale: evidence for the cross-method convergence of well-being measures. J Pers Assess. 1991 Aug;57(1):149-61. doi: 10.1207/s15327752jpa5701_17. PMID 1920028
- [Background] Nielsen MG, Ornbol E, Vestergaard M, Bech P, Larsen FB, Lasgaard M, Christensen KS. The construct validity of the Perceived Stress Scale. J Psychosom Res. 2016 May;84:22-30. doi: 10.1016/j.jpsychores.2016.03.009. Epub 2016 Mar 16. PMID 27095155